CLINICAL TRIAL: NCT06852209
Title: Cognitive Impairment Mechanisms and Training With Real Time-functional MRI Neurofeedback After Stroke
Brief Title: Training Cognition With Neurofeedback After Stroke
Acronym: CITRINeS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CHUBX 2023/43
Record Dates: First submitted 2024-12-02; First posted 2025-02-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Cognitive Impairment
Keywords: Stroke; Cognition; Real time-fMRI; Neurofeedback
MeSH Terms: conditions — Stroke; Cognitive Dysfunction | interventions — Neuropsychological Tests

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Training sessions of rt-fMRI NF. The experimental procedure will include four training sessions of rt-fMRI NF (1/week), preceded by a localizer session for the identification of the target networks, and followed by a tranfer session where the subjects will be asked to try to self-regulate their brain activity but without receiving feedback
  Interventions: Procedure: Cognitive remediation therapy; Procedure: Neuropsychological assessment; Procedure: Real-time functional MRI neurofeedack (rt-fMRI NF)
- Control group (Active Comparator): Four fMRI sessions but without receiving feedback
  Interventions: Procedure: Cognitive remediation therapy; Procedure: Neuropsychological assessment; Procedure: fMRI sessions

INTERVENTIONS:
Procedure: Cognitive remediation therapy — Cognitive remediation therapy as treatment as usual
Procedure: Neuropsychological assessment — Neuropsychological assessment to measure cognitive performances
Procedure: Real-time functional MRI neurofeedack (rt-fMRI NF) — Real-time functional MRI neurofeedack (rt-fMRI NF) is a procedure of brain-machine interface supporting self-regulation of brain activity, with promising results in the treatment of mental disorders. The main objective of the study is to evaluate in a pilot study, the ability of stroke patients to learn to self-regulate their brain activity in a priviledged direction.
  Arms: Experimental group
Procedure: fMRI sessions — fMRI sessions but without receiving feedback
  Arms: Control group

SUMMARY:
Post-stroke cognitive impairment (PSCI) is a common source of invisible disability. The actual techniques of cognitive remediation have been reported to have only a small effect, justifying the need to foster research in this field. Real-time functional MRI neurofeedack (rt-fMRI NF) is a procedure of brain-machine interface supporting self-regulation of brain activity, with promising results in the treatment of mental disorders. The main objective of the study is to evaluate in a pilot study, the ability of stroke patients to learn to self-regulate their brain activity in a priviledged direction, using rt-fMRI NF

DETAILED DESCRIPTION:
Stroke is a major source of cognitive impairment including slowdown of processing speed, executive functions disturbances, attention and memory loss, that can lead to invisible disability, even before the ultimate stage of dementia. The traditional techniques of cognitive remediation have been reported to have a small effect, and european scientific societies stated on the need to foster research in the field of PSCI, with the goal of preventing cognitive decline. PSCI mechanisms arising from functional MRI studies include a disconnexion of brain networks, with a loss of segregation between networks and integration within networks, centered on the frontoparietal network. Rt-fMRI NF is a psychophysiological procedure of brain-machine interface enabling to a subject to learn to self-regulate his brain activity in a desired direction, based on the brain haemodynamic response. Promising results in the treatment of mental disorders have been reported using rt-fMRI NF, but data are scarce in the field of cognitive rehabilitation after stroke. Based on the mechanisms of PSCI reported in fMRI studies, the goal of the present study is to evaluate the ability of stroke patients to learn to self-regulate a brain target using rt-fMRI NF. The brain target is defined by the difference of activation between the central executive network (CEN, or frontoparietal network) and the default mode network (DMN), known to be highly anticorrelated with the CEN in the healthy brain. The experimental procedure will include four training sessions of rt-fMRI NF (1/week), preceded by a localizer session for the identification of the target networks, and followed by a tranfer session where the subjects will be asked to try to self-regulate their brain activity but without receiving feedback. A control group will perform the four fMRI sessions but without receiving feedback. The two groups will receive cognitive remediation therapy as treatment as usual. Resting state scans and diffusion tensor imaging seqences will be performed before and after the intervention, to measure the changes in functional and structural connectivity. A neuropsychological assessment will be also performed before and after the intervention, to measure the changes in cognitive performances.

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* Right handed
* 18 ≤ years old < 75
* first-ever ischemic stroke on brain MRI in the past 3 to 6 months ;
* Persisting cognitive complaint 3 months after the ischemic stroke, proved by a MoCA score ≤ 26 (if educational level ≥ 12 years, or ≤ 25 if educational level < 12 years), and involving at least one of the following cognitive domains : executive functions, attention, and processing speed ;
* Ischemic stroke located in the territory of the middle cerebral artery and /or basal ganglia/thalamus ;
* NIHSS ≤ 5, without aphasia or severe visual disability empeding the understanding of the instructions, the neurofeedback task achievement, and/or the neuropsychological assessment ;
* No prestroke disability defined by a modified Rankin Scale ≤ 2 ;
* For women of childbearing potential, use of effective contraception and negative pregnancy test.
* Written informed consent by the patient.
* Coverage by the French Social Insurance

Exclusion Criteria:

* Previous cognitive impairment ;
* History of psychiatric disorder ;
* Current use of psychotropic medication ;
* MRI contraindication ;
* Pregnancy or breastfeeding ;
* Chronic disease empeding the follow-up of the subject during the lenght of the study ;
* Non fluently-French speakers ;
* Patient under legal protection.
* Patient unable of giving personal consent
* Emergency situation
* 1st MRI incomplete, not performed or not analyzable

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-10-28 (Estimated); Study Completion 2026-11-28 (Estimated)

PRIMARY OUTCOMES:
Differential CEN-DMN activity and imaging contrast between regulation and rest | Through study training completion, an average of 4 weeks
  Change from baseline to each training session on the CEN-DMN activity during regulation compared with rest, in the experimental and control groups

SECONDARY OUTCOMES:
Evolution of global cognition assessed by the Montreal Cognitive Assessment (MoCA) | Through study completion, an average of 6 weeks
  Change from baseline to the end of the study on the MoCA score. The MoCA score allows the detection of mild cognitive impairment and is ranged from 0 (minimum) to 30 (maximum : no cognitive impairment).
Evolution of executive functions assessed by a composite score | through study completion, an average of 6 weeks
  Change from baseline to the end of the study on a composite Z-score made from the averages of the Z-scores of the following tests :
  * verbal fluency : the subject is asked to cite a maximum of animals, letters starting with the letter P and V in 60 seconds) ;
  * memory span (working memory) : the subject is asked to restitute a maximum of the items of a list immediatly after hearing them) ;
  * Trail making Test (cognitive flexibility) : the subject is asked to link a set of digits in increasing order, alternating with letters, or items of different shapes or colors, the number of errors is recorded ;
  * Stroop task (inhibition capacity) : the subject is asked to name the font color of a list of words of colors which don't match their font color ;
  * Zoo testing plan (scheduling ability) : the subject is asked to follow a list of instructions for the visit of a zoo, while dealing with a list of constraints.
Evolution of attentional functions assessed by the Mesulam cancellation task | Through study completion, an average of 6weeks
  Change from baseline to the end of the study on the Mesulam cancellation task : the subject is asked to cancel a specific target among random arrays of structured and unstructured verbal and nonverbal stimuli.
Evolution of processing speed assessed by the Symbol Digit Modalities Test (SDMT) | Through study completion, an average of 6 weeks
  Change from baseline to the end of the study on the SDMT : the subject is provided with a set of symbols corresponding to numbers, and he is asked to write the symbols corresponding to a specific list of numbers in 5 minutes.
Evolution of memory functions assessed by the 16-item Free and Cued Recall | Through study completion, an average of 6 weeks
  Change from baseline to the end of the study on the 16-item Free and Cued Recall : the subject is asked to recall a set of 16 words presented by 4, immediately and after an interfering task, the number of free and cued correct recalls are recorded.
Evolution of visuospatial functions assessed by the Rey figure | Through study completion, an average of 6 weeks
  Change from baseline to the end of the study on the Rey figure : the subject is asked to copy a complex figure as quickly as possible, and then, to reproduce the figure without the model.
Evolution of language functions assessed byt the 40-item neuropsychological semantic battery | Through study completion, an average of 6 weeks
  Change from baseline to the end of the study on the 40-item neuropsychological semantic battery : the subject is asked to name a set of 40 living and non living items in verbal and visual conditions, across 6 subtests of matching.
Evolution of the Central Executive Network (CEN) activity | Through study training completion, an average of 4 weeks
  Change from baseline to each training session in the CEN activity recorded in the CEN mask during regulation compared with rest, in the experimental and control groups. The CEN mask is a binary mask individualized after running a pipeline for each subject, and the functional activity into this mask is extracted to assess the specific trajectory of the CEN activity.
Evolution of the Default Mode Network (DMN) activity | Through study training completion, an average of 4 weeks
  Change from baseline to each training session in the DMN activity recorded in the DMN mask during regulation compared with rest, in the experimental and control groups. The DMN mask is a binary mask individualized after running a pipeline for each subject, and the functional activity into this mask is extracted to assess the specific trajectory of DMN activity.
Evolution of activity in the whole brain | Through study training completion, an average of 4 weeks
  Change from baseline to each training session on the whole brain activity during regulation compared with rest, in the experimental and control groups
Evolution of resting state CEN and DMN activity | Through study completion, an average of 6 weeks
  Change in correlation between resting state CEN and DMN activity before intervention compared with after intervention.
Microstructural changes assessed by Fractional Anisotropy (FA) | Through study completion, an average of 6 weeks
  Change in median FA parameters before intervention compared with after intervention
Microstructural changes assessed by Mean Diffusivity (MD) | Through study completion, an average of 6 weeks
  Change in median MD parameters (mm2/sec) before intervention compared with after intervention
Microstructural changes assessed by Axial Diffusivity (AD) | Through study completion, an average of 6 weeks
  Change in median AD parameters (mm2/sec) before intervention compared with after intervention
Microstructural changes assessed by Radial Diffusivity (RD) | Through study completion, an average of 6 weeks
  Change in median RD parameters (mm2/sec) before intervention compared with after intervention
Differential CEN-DMN activity and imaging contrast between regulation and rest, without neurofeedback | Through study completion, an average of 6 weeks
  Change from baseline to the last fMRI session (" transfert session " without neurofeedback) on the CEN-DMN activity during regulation compared with rest, in the experimental and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila SAGNIER, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France